CLINICAL TRIAL: NCT00932399
Title: Weight Change, Physical Activity and Health Promotion in Veteran Amputees
Brief Title: Longitudinal Study of Weight Change Following Lower Limb Amputation
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: F6982-W
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Amputation Wound; Traumatic Amputation of Toe; Dysvascular Amputation of Lower Limb

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Underwent a procedure at a VA medical facility in VISN 20 for a lower limb amputation between 1997 and 2008
- Group 2: No history of lower limb amputation

SUMMARY:
The purpose of this study is to assess weight change in a population of Veterans with amputations. Little is known about the how weight changes following an amputation. It is widely believed that many patients experience weight gain following amputation. This study aims to identify magnitude of weight changes following amputation and determine characteristics associated with weight gain. Information on weight change trajectories would be useful to better understand long-term health consequences associated with amputation and to design and target interventions to encourage weight maintenance and general health promotion for groups at high risk of weight gain.

ELIGIBILITY:
Inclusion Criteria:

"Exposed" cohort:

* incident lower limb amputation during the study period (1/1997-12/2008) in VISN 20
* >= 1 plausible weight recoded in the medical record at baseline (defined as 8 weeks before amputation or 2-8 weeks post amputation)
* >=1 weight measured post amputation (2 months to 42 months post amputation)

"Unexposed" (comparison) cohort:

* no lower limb amputation during the study period
* no prior history of amputation
* >= 2 plausible recorded weights including at least one in the 2-6 weeks after their reference date ("baseline").
* Alive at least 18 months after "baseline"

Exclusion Criteria:

* female (due to small number of women with lower limb amputations)
* lack information on any of the characteristics used for matching (e.g., birth year/age and height to calculate body mass index)

Ages: 27 Years to 89 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans who received care at a VISN20 medical facility between 1997 and 2008
Sampling Method: Probability Sample
Enrollment: 4549 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alyson J. Littman, PhD MPH, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

REFERENCES:
- [Result] Bouldin ED, Thompson ML, Boyko EJ, Morgenroth DC, Littman AJ. Weight Change Trajectories After Incident Lower-Limb Amputation. Arch Phys Med Rehabil. 2016 Jan;97(1):1-7.e1. doi: 10.1016/j.apmr.2015.09.017. Epub 2015 Oct 8. PMID 26453769

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Underwent a procedure at a VA medical facility in Veterans Integrated Service Network #20 for a lower limb amputation between 1997 and 2008
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 759 | 3790
Completed | 759 | 3790
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 759 | 3790 | 4549
Age, Customized [Number; unit: participants]
  <55 years | 141 | 705 | 846
  55-64 years | 294 | 1470 | 1764
  65-74 years | 200 | 995 | 1195
  75-89 years | 124 | 620 | 744
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 759 | 3790 | 4549

OUTCOME MEASURES:

1. Primary Outcome: % Weight Change From Baseline
Description: Time window for 3 years is 31-39 months after baseline
Time Frame: At ~3 years after baseline
Measure: Mean (95% Confidence Interval); unit: % weight change
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 759 | 3790
% weight change | 5.5 [4.1 to 6.9] | 0.9 [0 to 1.8]

ADVERSE EVENTS:
Description: Serious and other [non-serious] adverse events were not collected or assessed as part of the study. This was a retrospective study using medical records.
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No